CLINICAL TRIAL: NCT07004270
Title: Evaluation of the Impact of Emergency Advanced Practice Nurses One Year After Implementation in the Adult Emergency Department of a French University Hospital - A Monocentric Cross-sectional Observational Study
Brief Title: Evaluation of the Impact of Emergency Advanced Practice Nurses One Year After Implementation in the Adult Emergency Department of a French University Hospital
Acronym: IMPACTED
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IMPACTED
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Advanced Practice Nursing; Emergency Departments; Patient Satisfaction
MeSH Terms: conditions — Emergencies; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In France and around the world, emergency care facilities are facing increasing demand, with rising waiting times. Differentiating care pathways, notably by opening a fast-track unit, helps to improve patient flow and waiting time; which contributes to patient satisfaction. However, a link between patient satisfaction and waiting time is not always found when patients perceive a humanistic approach in care.

The implementation of an advanced practice nurse in an emergency department is a way to graduate the offer of care and reduce waiting times before consultation and length of stay for patients with minor degree of severity. In this care context, Advanced Practice Nurses maintain and even improve patient satisfaction.

Since July 2024, two Advanced Practice Nurses have integrated Poitiers University Hospital's adult emergency department. Considering the existing and ongoing literature to knowledge, an evaluation of the impact of emergency Advanced Practice Nurses 1 year after their implementation in a French University Hospital would be the first study of its kind.

According to the results of previous international studies, the investigators assume that emergency Advanced Practice Nurses activities have a positive impact on the French healthcare system: on the quality of care perceived by patients and on the emergency care pathways of all fast-track patients by maintaining the same level of safety. This study aims to evaluate the impact of emergency Advanced Practice Nurses in a French University Hospital on patient perception of quality of care, safety and patient care pathways in emergency departments.

This monocentric cross-sectional observational study is a prospective survey of patient satisfaction and experience with a satisfaction questionnaire; and a retrospective survey on routine care data.

The study's main objective is to evaluate the impact of emergency Advanced Practice Nurses in a French University Hospital on patient-perceived quality of care by measuring the overall satisfaction of patients who receive care from Advanced Practice Nurses during their emergency care pathway. Overall patient satisfaction will be measured in a survey conducted with a patient satisfaction and experience questionnaire.

The secondary objectives of this study are several:

* Assess patients' acceptability of being cared by an emergency Advanced Practice Nurse
* Evaluate patient satisfaction with the communication and care relationship with an emergency Advanced Practice Nurse
* Evaluate the rate of recommendation of an emergency Advanced Practice Nurse by the patients who receive care from an Advanced Practice Nurse
* Evaluate the safety of care pathways including an emergency Advanced Practice Nurse
* Evaluate the impact of emergency Advanced Practice Nurses implementation on emergency care pathways for fast-track patients

Consistent with each objective and outcome, the study will compare:

* groups before and after the implementation of emergency Advanced Practice Nurses
* or subgroups in the period after implementation of advanced practice nurses: with and without emergency Advanced Practice Nurses intervention The anonymous patient satisfaction and experience survey will be sent by a link in a verified e-mail during the emergency department visit of patients included in the study, admitted to emergency department between 02/06/2025 and 29/06/2025.

Routine care data will be collected from Poitiers hospital medical records for fast-track patients who did not refuse to take part in the study during the following periods:

* Before Advanced Practice Nurses' implementation from 05/27/2024 to 06/23/2024
* After Advanced Practice Nurses' implementation from 02/06/2025 to 29/06/2025

ELIGIBILITY:
Inclusion Criteria:

* Patient arrived in fast-track unit during Advanced Practice Nurses' attendance periods
* Adult over or equal 18 years old

Exclusion Criteria:

* Patient who refused to participate to the research
* Patient deprived of total or partial liberty by a judicial or administrative decision
* Patients under guardianship or trusteeship
* Patient with diagnosed cognitive disorders
* Non-French-speaking patient
* Patients who left without waiting for treatment or against medical advice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen in the fast-track emergency department during the inclusion periods, who were cared by an Advanced Practice Nurse or physician, and who did not refuse to be included in the study by gathering their routine care data and, if applicable, their anonymous responses to the patient satisfaction survey.
Sampling Method: Non-Probability Sample
Enrollment: 921 (Actual)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Compare rate of patients overall satisfied of care received in the emergency department with Advanced Practice Nurse's intervention to the overall satisfaction rate without Advanced Practice Nurse's intervention | Day 1

SECONDARY OUTCOMES:
Rate of patients who have refused care from an emergency Advanced Practice Nurse | Day 1
Rate of patients satisfied with the clearness of information and/or responses about their health and cares | Day 1
Rate of patients satisfied with the relation with the health providers | Day 1
Rate of patients reinsured after an emergency visit | Day 1
Rate of patients who would recommend emergency care by an Advanced Practice Nurse | Day 1
Compare rates of 72-hours reconsultation in emergency departments for the same reason, of fast-track patients care pathway with and without Advanced Practice Nurse's intervention | Day 3
Compare rates of complaints related to patients fast-track care in pathway with and without Advanced Practice Nurse's intervention | Day 1
Compare rates of adverse events and serious adverse events for patients in the fast-track pathway with and without Advanced Practice Nurse | Day 1
Compare waiting times in minutes before first medical contact or with Advanced Practice Nurse in the fast-track pathway before and after Advanced Practice Nurses' implementation | Day 1
Compare median length of stay of fast-track patient's pathway before and after Advanced Practice Nurses' implementation | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Poitiers, Poitiers, France, France